CLINICAL TRIAL: NCT00630448
Title: Collection of Blood in Normal Subjects and Subjects With Von Willebrand Disease (VWD)
Status: Withdrawn | Type: Observational
Why Stopped: Prinicipal Investigator initiated study closure.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0708009371
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Control Group. Normal (healthy) individuals without Von Willebrand Disease.
- Group 2: Case Group. Individuals with known Von Willebrand Disease.

SUMMARY:
Von Willebrand disease is an inherited bleeding disorder that impacts the blood's ability to clot properly. Von Willebrand disease is cause by the lack or not working substance in the blood known as Von Willebrand factor.

Current therapy for Von Willebrand disease includes desmopressin acetate (DDAVP) and /or VWF/FVIII concentrates. Patients with severe Von Willebrand disease face a lifetime of weekly treatments and mounting medical bills. Gene therapy could help these patients improve their quality of life by providing the missing factors necessary for the blood's ability to clot properly.

The gene transfer options being studied include naked DNA, viral gene transfer vectors encoding Von Willebrand factor transgenes, and ex vivo cell therapy. The latter involves transplantation of the patient's own cells modified with a corrected copy of the defective gene. Human blood outgrowth endothelial cells (BOEC) display all the properties needed for successful ex vivo cell therapy. We plan to obtain blood samples from normal research subjects and patients with Von Willebrand Disease in order to isolate blood outgrowth endothelial cells (BOEC) from peripheral blood, and develop a ex vivo gene therapy for Von Willebrand Disease.

DETAILED DESCRIPTION:
Aim: The purpose of this protocol is to obtain blood samples from normal research subjects and patients with Von Willebrand disease in order to isolate blood outgrowth endothelial cells (BOEC) from peripheral blood, and develop a ex vivo gene transfer for Von Willebrand disease.

Experimental procedure. This protocol is designed to gather approximately 90 ml (6 tablespoons) of blood from normal individuals without Von Willebrand disease and individuals with known Von Willebrand disease. A total of 20 normal individuals and 20 Von Willebrand disease patients will be enrolled into the study.

Studies to be performed on the blood samples:

Each blood draw will require 10 large blue/black capped (Na Citrate) vacutainer (16x125mm, BD# 362761, Cell Preparation Tubes (CPT) to be filled from each volunteer. All the blood will be used for cell processing.

In initial proof-of-concept experiments, BOEC lines will be established from the peripheral blood of normal individuals and research subjects with Von Willebrand disease. Following culture and phenotypic characterization, they will be transduced with a lentivirus gene transfer vector expressing a reporter gene or wild-type Von Willebrand factor. After demonstrating successful transduction, the next step will be to write an animal protocol that will introduce the modified cells into immunocompromised mice and monitor the mice for stable implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Normal subjects:

   - study individuals will be taken from those enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"
2. Subjects with von Willebrand Disease

   * a definitive diagnosis on VWD from a patient's physician
   * all subjects should be able to provide informed consent
   * males or females 18-70 years of age

Exclusion Criteria:

1. Normal individuals

   * individuals with a history of bleeding disorders
   * individuals with anemia (defined as females with an Hgb concentration less than 12 and males with an HgB concentration less than 12.5)
2. Subjects with VWD

   * females who are pregnant will not be accepted into the study
   * individuals with anemia (defined as females with an Hgb concentration less than 12 and males with an Hgb concentration less than 12.5)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Source of subjects will be the population of individuals with known Von Willebrand Disease and the normal population from protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Blood outgrowth endothelial cells from peripheral blood | Through study completion, an average of 1 month
  The number of isolated blood outgrowth endothelial cells from peripheral blood will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No